CLINICAL TRIAL: NCT00143442
Title: A 5-Week, Randomized, Double-Blind, Placebo-Controlled Multi-Center Study Of [S,S]-Reboxetine In Patients With Postherpetic Neuralgia (PHN), Who Are Gabapentin Treatment Failures.
Brief Title: Study of [S,S]-Reboxetine in Patients With Postherpetic Neuralgia, Who Are Gabapentin Treatment Failures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061001
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2006-08-08 (Estimated); Status verified 2006-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
The purpose of this study is to determine the effectiveness of [S,S]-Reboxetine in the treatment of chronic pain following a shingles infection in patients who are Gabapentin treatment failures.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after the healing of shingles skin rash.
* Patients at screening must have a score > or = 40 mm on the pain visual analogue scale.

Exclusion Criteria:

* Patients with poor renal function.
* Patients with other severe pain, that may impair the self-assessment of the pain due to shingles.
* Patients with abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184
Dates: Start 2003-12; Study Completion 2004-10

PRIMARY OUTCOMES:
The numerical pain intensity rating scale is used to assess pain and a change from baseline in pain score for week 5 will be calculated.

SECONDARY OUTCOMES:
- The mean endpoint (week 5) sleep interference score change from baseline - Analysis of the Patient Global Impression of Change - Analysis of the Clinical Global Impression of Change - Analysis of the SF-McGill questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer